CLINICAL TRIAL: NCT02821481
Title: The Interactive Effects Of Beta-Alanine Supplementation and Resistance Training on Muscular Endurance in Older Adults
Brief Title: Beta-alanine and Elder Endurance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20140412
Record Dates: First submitted 2016-06-28; First posted 2016-07-01 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Physical Endurance
Keywords: Neuromuscular; Supplementation; Elderly
MeSH Terms: interventions — beta-Alanine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Beta-alanine and muscular endurance exercise (Experimental): Receive 3.2 g/day beta-alanine and 3 days per week of endurance resistance training for 12 weeks
  Interventions: Dietary Supplement: Beta-alanine; Behavioral: Muscular endurance exercise
- Beta-alanine without muscular endurance training (Experimental): Receive 3.2 g/day beta-alanine with no endurance resistance training for 12 weeks
  Interventions: Dietary Supplement: Beta-alanine
- Placebo and muscular endurance exercise (Placebo Comparator): Receive similar dextrose placebo and 3 days per week of endurance resistance training for 12 weeks
  Interventions: Dietary Supplement: Placebo; Behavioral: Muscular endurance exercise
- Placebo without muscular endurance training (Placebo Comparator): Receive similar dextrose placebo with no endurance resistance training for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Beta-alanine
  Arms: Beta-alanine and muscular endurance exercise; Beta-alanine without muscular endurance training
Dietary Supplement: Placebo
  Arms: Placebo and muscular endurance exercise; Placebo without muscular endurance training
Behavioral: Muscular endurance exercise
  Arms: Beta-alanine and muscular endurance exercise; Placebo and muscular endurance exercise

SUMMARY:
The purpose for this study is to determine if beta-alanine supplementation combined with endurance-based resistance training can increase gains in muscular endurance to a greater extent than endurance-based resistance-training alone in older adults.

ELIGIBILITY:
Inclusion Criteria:

* 60-90 years of age
* Living independently (not residing in an assisted living facility)
* Through testing are found not to have sarcopenia
* Gait speed > 1 m/s
* Skeletal Muscle Index > 37% in men and > 27.6 % in women
* Exclusion Criteria
* Responding with a "yes" to any question on the PAR-Q.
* Are currently pregnant, or plan to try and become pregnant during the study
* Functional impairments that could impede the person's ability to participate in a resistance training program
* Current or recent use of supplements (within the past 3 months for non-alanine containing supplements or one year for supplements containing beta-alanine). Individuals taking only basic multivitamins (without any herbal co-ingredients) may still be allowed to participate. These situations will be reviewed on a case-by-case basis.
* Are currently enrolled in a regular exercise program (more than once per week)
* Current or recent smoker
* Use of medication containing corticosteroids
* Mini-mental score of 21 or below
* Severe musculoskeletal impairment
* Uncontrolled chronic disease
* Major depression
* Severe vestibular problems

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Performance of Daily Activities | baseline, 12 weeks
  Short Physical Functional Performance test

SECONDARY OUTCOMES:
Change in Body Fat | baseline, 12 weeks
  Body fat assessment via bioimpedance
Change in Muscular Endurance | baseline, 12 weeks
  20 repetitions to measure decline in muscular power across repetitions
Change in Muscular Strength | baseline, 12 weeks
  Maximal weight that could be lifted one time (1RM)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F. Signorile, PhD, Principal Investigator — University of Miami
Locations (1):
- Max Orovitz Laboratories, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No